CLINICAL TRIAL: NCT04685629
Title: Long-term Follow-up of Covid-19 Patients in Their Home Environment After Hospitalization in a Covid Department or Intensive Care Unit
Brief Title: Covid-19 Long-term Revalidation Follow-up
Acronym: Colonel
Status: Withdrawn | Type: Observational
Why Stopped: failed to included during covid pandemic
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Davina Wildemeersch, MD, University Hospital, Antwerp
Other Study IDs: Colonel
Record Dates: First submitted 2020-12-21; First posted 2020-12-28 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Covid19
Keywords: COLONEL; Tele-monitoring
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 25 post ICU-patients — patients who were hospitalized in an intensive care unit
Other: 25 post non-ICU patients — patients who were not hospitalized in an intensive care unit

SUMMARY:
In this monocentric, prospective and descriptive trial we want to evaluate the long-term consequences for patients treated for Covid-19. Covid patients who were hospitalized for min. 5 days either in a Covid-19 department or in intensive care unit will be followed-up for 8 weeks after hospital discharge. This is done via an innovative electronic platform in the home environment (UZA@home). On the one hand the quality of life, rehabilitation and reintegration of the patient will be evaluated and on the other hand the patient will be screened for various psychosocial aspects such as anxiety, depression and post-traumatic stress syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Adult age
* Hospitalization with proven Covid-19 infection with a minimum stay of 5 days
* Signed Informed Consent

Exclusion Criteria:

* The patient does not have a smartphone or computer with internet connection.The patient is not sufficiently skilled in entering data via a digital interface. This degree of skill is estimated by the research doctor or nurse.
* Patient in a palliative setting (DNR 2 or higher outside of COVID condition
* The patient does not speak the Dutch language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We want to follow up 50 patients from hospital discharge, where we want to distinguish 2 groups:
  * patients after admission to the intensive care unit (25)
  * patients without admission to the intensive care unit (25)
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-05-07 (Actual); Primary Completion 2022-05-22 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Health related Quality of life (general well-being) questionnaire | in the first 7 days after hospital discharge
  Evaluation of Quality of Life after hospitalization due to COVID-19 infection using the EQ-5D-5L questionnaire
Health related Quality of life (general well-being) questionnaire | 4 weeks after hospital discharge
  Evaluation of Quality of Life after hospitalization due to COVID-19 infection using the EQ-5D-5L questionnaire
Health related Quality of life (general well-being) questionnaire | 8 weeks after hospital discharge
  Evaluation of Quality of Life after hospitalization due to COVID-19 infection using the EQ-5D-5L questionnaire

SECONDARY OUTCOMES:
Revalidation & Reintegration | daily, up to 8 weeks after hospital discharge
  Evaluation of revalidation of the patient after hospitalization (daily functioning and mobilization via a daily diary and objective measurements by means of remote monitoring techniques (saturation measurement, activity tracker, sleep monitor)).
Depression and/or anxiety | 3 times after hospital discharge: first at week 0, second time at week 4, third time 8 weeks after discharge
  Evaluation of depression and anxiety of the patient after hospitalization via the HADS (Hospital Anxiety and Depression Scale) questionnaire
Post traumatic stress syndrome | 8 weeks after hospital discharge
  Evaluation of post traumatic stress syndrome of the patient after hospitalization via the PTSS questionnaire (of Erik De Soir)

CONTACTS AND LOCATIONS:
Locations (1):
- Antwerp University Hospital, Edegem, Antwerpen, Belgium